CLINICAL TRIAL: NCT01312948
Title: Pediatric Nasal Mask (Pixi) Usability Study
Brief Title: Study of the Usability and Efficacy of a New Pediatric CPAP Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA13122010
Record Dates: First submitted 2011-02-06; First posted 2011-03-11 (Estimated); Results first posted 2012-03-19 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Obstructive Sleep Apnea; Respiratory Insufficiency
Keywords: Obstructive sleep apnea; OSA; CPAP; CPAP mask; Non-invasive ventilation; NIV
MeSH Terms: conditions — Sleep Apnea, Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prototype mask (Experimental)
  Interventions: Device: Prototype mask (known as Pixi)

INTERVENTIONS:
Device: Prototype mask (known as Pixi) — This is a prototype mask to be used with continuous positive airway pressure (CPAP) or non-invasive ventilation (NIV) therapy. The mask attaches to the face, covering the nose, and is kept in place with headgear. Therapy is delivered through the mask via a tube which attaches to the CPAP or NIV device.
  Other Names: ResMed Pixi paediatric mask

SUMMARY:
This study will evaluate a newly developed pediatric mask (known as Pixi) on children aged 2-7 using continuous positive airway pressure (CPAP), or Non-invasive ventilation (NIV) treatment. The participants will undergo a monitored sleep study, followed by a 7 night trial of the Pixi mask in the home environment. During the study usability will be measured through questionnaires filled in by the parent and clinician.

The study hypothesis is that the usability of the mask will be superior to the patient's usual mask.

DETAILED DESCRIPTION:
This is a prospective, single group, un-blinded study sponsored by ResMed Ltd to investigate the usability of the ResMed Pediatric Nasal Mask (Pixi).

Patients will be recruited from the study site's database. Parents/ guardians of patients who meet the selection criteria and voluntarily agree to participate in the study will be approached by the investigative team to obtain informed consent.

Patients will attend the clinic where baseline information will be collected, including information about the patient's current therapy and data from their last PSG study. Information will be recorded on case report forms (CRF's). Data from the patient's current device will be downloaded during this visit. At this time the Pixi mask will be fitted and adjusted until it is comfortable for the child. The patient's device will be switched to a ResMed VPAP III ST-A with QuickNav if they are not already using one. The VPAP III ST-A with QuickNav will be used in the same mode (CPAP or Bi-level) as the patient's current device.

The participants will undergo a monitored PSG study on the first night of the trial. They will use the Pixi mask and the VPAP III ST-A with QuickNav during this PSG. The initial therapy settings will be based on the child's usual therapy, with any therapy setting modifications made as clinically required during the PSG.

Patients will then use the Pixi mask with the VPAP III ST-A with QuickNav in the home environment for 7 nights. After using the mask in the home environment, the child's legal guardian will rate their satisfaction with the Pixi mask as compared to the child's current mask. The child will also be asked to evaluate the mask if they are able.

ELIGIBILITY:
Inclusion Criteria:

* Is between 2-7 years of age
* Is a current PAP (Bi-level or CPAP) therapy user, defined as being on PAP therapy for at least 1 month prior to study entry
* Is a current user of a nasal mask
* Legal guardian can read and comprehend English
* Legal guardian is willing to give written informed consent

Exclusion Criteria:

* Recent sinus surgery (within 6 weeks of study entry)
* Concurrent participation in other clinical trials
* History of clinically significant epistaxis in the past 6 months
* Known co-morbidities that, per clinical judgment, would prevent compliance to therapy
* Other reasons for non-compliance that affect subject's ability to use therapy such as primary claustrophobia
* Significant cardiac disease

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret-Anne Harris, MBBS, FRACP, Principal Investigator — Lady Cilento Children's Hospital, Brisbane
Locations (1):
- Mater Children's Hospital, Brisbane, Queensland, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Mater Children's Hospital patient database. Patients were recruited from January - April 2011. Participants attended Mater Children's Hospital Sleep Unit to take part in the study
Groups:
- Prototype Mask: New paediatric mask system (Pixi) designed for children aged 2-7 years using Positive airway pressure (PAP) therapy
Period: Overall Study
Arm/Group | Prototype Mask
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prototype Mask
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.6 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  Australia | 6

OUTCOME MEASURES:

1. Primary Outcome: Usability Ratings of the Pixi Paediatric Mask Compared With the Child's Current Mask
Description: Before trialling the Pixi mask, parents rated the usability of their child's usual mask using a 0-10 Likert Scale where 0 = poor and 10 = excellent. After trialling the Pixi mask, parents then completed the same questionnarie for the Pixi mask.
  Usability was defined as a single overall score of mask performance. Parents considered mask seal, comfort, stability and red marks when scoring each mask for usability.
Time Frame: 8 nights use
Population: Analysis was as per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pixi Paediatric Mask Usability: Usability (overall performance) score of the Pixi paediatric mask
- Usual Mask: Usability (overall performance) score of the child's usual CPAP mask
Arm/Group | Pixi Paediatric Mask Usability | Usual Mask
Number analyzed (Participants) | 6 | 6
units on a scale | 7.17 (2.93) | 5.83 (1.94)

2. Secondary Outcome: Equivalence of Apnea-hypopnea Index (AHI) on the New Pixi Mask Compared With the Child's Usual Mask
Description: Apnea-Hypopnea index (AHI) is a measure of the severity of sleep disordered breathing (SDB). It describes how many events of compromised breathing occur each hour of sleep. The higher the AHI, the more severe the SDB (mild 5-15, moderate 15-30, severe >30). In clinical practice an AHI <5 demonstrates efficacy of treatment. AHI was recorded during a monitored sleep study on the new Pixi mask, and compared with the AHI from a monitored sleep study on the child's usual mask. The outcome hypothesis was that the Pixi mask AHI would be equivalent or reduced compared to the patients usual mask
Time Frame: >4 hours monitored sleep study
Population: Analysis was as per protocol
Measure: Mean (Standard Deviation); unit: apnea hypopnoea index
Groups:
- Pixi Paediatric Mask: Apnea hypopnoea index from a monitored sleep study of the new Pixi mask. An apnea hypopnoea index of <5 demonstrates treatment efficacy
- Usual Mask: Apnea hypopnoea index from a monitored sleep study of the child's usual CPAP mask. An apnea hypopnoea index of <5 demonstrates treatment efficacy
Arm/Group | Pixi Paediatric Mask | Usual Mask
Number analyzed (Participants) | 6 | 6
apnea hypopnoea index | 0.85 (0.76) | 3.25 (1.57)

ADVERSE EVENTS:
Arm/Group | Prototype Mask
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No